CLINICAL TRIAL: NCT06259214
Title: Aesthetic Efficacy of Resin Infiltration Using Different Conditioning Methods: 24-Month Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Dr Emel Karaman, Assoc.Prof. Emel Karaman, Ondokuz Mayıs University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1700213
Record Dates: First submitted 2024-01-29; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: White Spot Lesion
Keywords: Color stability; Fluorescence; Resin infiltration; White spot lesion
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- regular brushing (No Intervention): regular brushing
- 15% HCl gel (Active Comparator): 15% HCl gel (Icon Etch, DMG, Hamburg, Germany) was applied to the WSLs for 2 min, followed by water rinsing and drying with compressed air (each for 30 s)
  Interventions: Other: 15% HCl gel
- 37% H3PO4 gel (Active Comparator): 37% H3PO4 gel (Scotchbond Etchant, 3M ESPE, St. Paul, MN, USA) was applied to the WSLs for 30 s, which were then water rinsed and dried with compressed air (each for 30 s)
  Interventions: Other: H3PO4 gel
- Er:YAG laser (Active Comparator): Er:YAG laser (Fotona AT Fidelis III, Ljubljana, Slovenia) was applied for 10 s with the following operating parameters: energy 300 mJ, frequency 10 Hz, wavelength 2.94 μm, short pulses of 10 pulses per second, pulse time 180 ms, distance 1 mm away from lesion, water spray cooling 80%.
  Interventions: Other: Er:YAG laser

INTERVENTIONS:
Other: 15% HCl gel — Icon , DMG, Hamburg, Germany
  Arms: 15% HCl gel
Other: H3PO4 gel — Scotchbond Etchant, 3M ESPE, St. Paul, MN, USA
  Arms: 37% H3PO4 gel
Other: Er:YAG laser — Fotona AT Fidelis III, Ljubljana, Slovenia
  Arms: Er:YAG laser

SUMMARY:
Objective: To assess color and fluorescence changes in white spot lesions (WSLs) using different surface conditioning methods prior to resin infiltration: 24-months follow-up Methods: Thirty patients with each at minimum four WSLs after bracket debonding were included. After baseline fluorescence and color measurements, the lesions were randomly divided into four groups (n = 30): G1 (control): regular brushing, G2: 15% HCl gel (Icon Etch), G3: 37% H3PO4 gel (Scotchbond Etchant), G4: Er:YAG laser (Fotona AT Fidelis III). The lesions were desiccated with Icon Dry and then Icon Infiltrant (DMG) was applied. In the treatment groups, color and fluorescence were examined at baseline (T0), just after the resin infiltration treatment (T1), and after 6 (T2) and 24 months (T3). In the control group, the examinations were performed at baseline (T0) and after 6 (T2) and 24 months (T3).

DETAILED DESCRIPTION:
Prior to the study an experienced investigator (EK) attended a training and calibration session (k value = 0.88) and evaluated the severity of WSLs under direct illumination using a dental lamp with the aid of a standard 3.0× loupe (Keeler, Windsor, UK). Isolation was achieved with a cotton roll and suction. For the visual severity evaluation, all teeth were cleaned and air dried for 5 s and each lesion was scored according to ICDAS II free smooth-surface criteria [20]. Lesions with code 1 (first visual change after prolonged air drying) and code 2 (distinct visual changes without air drying) were included. The teeth were cleaned with a rubber cup and pumice, rinsed, and air dried (each for 30 s).

The same investigator (EK) used a DIAGNOdent Pen 2190 (Kavo, Biberach, Germany) to score each lesion afterwards. Before every scoring session, the device was calibrated using the standard ceramic according to the manufacturer's instructions. The teeth were rinsed and air dried before registration and a type B probe tip was positioned on the buccal surface of the tooth and rotated around its vertical axis until the peak reading was displayed on the panel. All measurements were taken 3 times and the average fluorescence value was recorded.

Out of 40 consecutive patients between 14 and 21 years of age who had just finished their fixed orthodontic treatment, 4 patients declined to participate in the trial and 6 patients did not meet the inclusion criteria, and 30 patients (18 females, 12 males, aged 15-19 years, mean age 17.1 years) with at least four WSLs on the buccal surfaces after bracket debonding were included in the trial. Patients with any systemic disease, bad oral hygiene, a smoking habit, enamel hypoplasia, staining, fluorosis, or restoration or cavity in any teeth with WSLs were excluded from the study. At the end of the clinical examination a total of 120 non-cavitated, unrestored WSLs after multibracket treatment on the buccal surfaces of the anterior and premolar teeth in the upper and lower jaws of 30 patients were included.

A spectrophotometer (SpectroShade; Medical High Technologies, Italy) was used to measure color parameters in the same examination room with standardized light conditions. The spectrophotometer was calibrated before the measurements of each specimen using a standard white background. The mouth piece attached to the intraoral camera of the spectrophotometer was placed at 90° on the alveolar process above each tooth. After correct placement of the optic handpiece, the examiner checked that the tooth appeared in the center of the yellow target box on the computer screen, and the opposing teeth, the tongue, and lips were not visible on the screen. The results from each tooth obtained by spectrophotometer were recorded, with the mean values of L*, a*, and b* automatically calculated at three consecutive times by positioning the intraoral camera, removing it, and then repositioning it. Three consecutive readings were taken using the spectrophotometer and the mean values were recorded.

Treatment

After rubber dam placement, the lesions of each patient were randomly divided into 4 groups (n = 30):

G1 (control): The control group received no treatment except regular brushing, G2: 15% HCl gel (Icon Etch, DMG, Hamburg, Germany) was applied to the WSLs for 2 min, followed by water rinsing and drying with compressed air (each for 30 s).

G3: 37% H3PO4 gel (Scotchbond Etchant, 3M ESPE, St. Paul, MN, USA) was applied to the WSLs for 30 s, which were then water rinsed and dried with compressed air (each for 30 s).

G4: An Er:YAG laser (Fotona AT Fidelis III, Ljubljana, Slovenia) was applied for 10 s with the following operating parameters: energy 300 mJ, frequency 10 Hz, wavelength 2.94 μm, short pulses of 10 pulses per second, pulse time 180 ms, distance 1 mm away from lesion, water spray cooling 80%.

The lesions were desiccated with ethanol (Icon Dry, DMG, Hamburg, Germany) and air dried for 30 s. Then resin infiltrant (Icon Infiltrant, DMG, Hamburg, Germany) was applied to the tooth surface and allowed to penetrate for 3 min. A cotton roll was used to wipe excess material from the surface, and the material then was light cured for 40 s with an LED device (EliparTM S10; 3M ESPE, St. Paul, MN, USA) with 1200 mW/cm2 light intensity in standard continuous mode. The clinician repeated the infiltration step for 1 min to infiltrate any remaining porosities. Dental floss was used to remove any excess resin from the proximal areas. Then polishing was conducted with Sof-Lex disks (3M ESPE, St. Paul, MN, USA) using a slow-speed handpiece. The disks were used in a decreasing sequence of granulation and each disk was used for 5 s. The same clinician (KAU) conducted all restorative procedures.

All patients were given oral hygiene instructions and oral hygiene packages, which included a toothbrush (Oral B, Advantage Sensitive, P&G Oral Health Care, Mason, OH, USA), fluoride toothpaste (Pro-Expert Professional Protection, Ipana, Gross-Gerau, Germany), and dental floss (Oral B, Essential floss, P&G Oral Health Care, Mason, OH, USA). The patients were asked not to use any other dental products during the study period and the oral hygiene packages were renewed every 2 months.

Follow up examination All patients attended the follow-up visits. New caries formation was evaluated during the follow-ups. In the treatment groups the DIAGNOdent Pen and spectrophotometer examinations were performed at baseline (T0), just after the resin infiltration treatment (T1), and after 6 (T2) and 24 months (T3). In the control group, the DIAGNOdent Pen and spectrophotometer examinations were performed at baseline (T0) and after 6 (T2) and 24 months (T3). Fluorescence and color values were recorded as previously described by the same investigator (EK), who was blinded regarding the treatment group allocation of the teeth.

The differences in fluorescence and color values were evaluated by taking into account the differences between the initial values and the values at the different evaluation times. L*, a*, and b* were measured each time, and the changes in them (ΔL, Δa, and Δb) were calculated. The L*-axis indicates how light a sample is (0 is black and 100 is white). The red/green axis is represented by the a*-value, with an increase meaning a higher red color component. The yellow/blue axis is represented by the b*-value, with an increase meaning higher yellow color. The color change ΔE<3.7 is considered a clinically acceptable color difference [9] and ΔE for each tooth was calculated as follows:

ΔE= [(ΔL)2+ (Δa)2+ (Δb)2]1/2 Statistical analysis The normality of the variables was evaluated with the Kolmogorov-Smirnov test and the homogeneity of the variances was evaluated with the Levene test. Variables were summarized as median [25th-75th percentile] values. In the variables that met the parametric test assumptions, the differences between groups and within groups were tested with analysis of variance in repeated measurements. The Bonferroni test was used for pairwise comparisons. In the variables that did not meet the parametric test assumptions, the differences between the groups were determined with the Friedman test and the differences between the groups were determined with the Kruskal-Wallis test. In the event of a difference, pairwise comparisons were conducted with Dunn's test.

ELIGIBILITY:
Inclusion Criteria:

at least four white spot lesions on the buccal surfaces after bracket debonding

Exclusion Criteria:

any systemic disease bad oral hygiene smoking habit enamel hypoplasia staining fluorosis restoration or cavity in any teeth with white spot lesions

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2019-01-06 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
color change | 24 month
  A spectrophotometer (SpectroShade; Medical High Technologies, Italy) was used to measure color parameters. The spectrophotometer was calibrated before the measurements of each specimen using a standard white background. The mouth piece attached to the intraoral camera of the spectrophotometer was placed at 90° on the alveolar process above each tooth. After correct placement of the optic handpiece, the examiner checked that the tooth appeared in the center of the yellow target box on the computer screen, and the opposing teeth, the tongue, and lips were not visible on the screen. The results from each tooth obtained by spectrophotometer were recorded, with the mean values of L*, a*, and b* automatically calculated at three consecutive times by positioning the intraoral camera, removing it, and then repositioning it. Three consecutive readings were taken using the spectrophotometer and the mean values were recorded.Higher values indicate more color change.
fluorescence loss | 24 monrth
  DIAGNOdent Pen 2190 (Kavo, Biberach, Germany) was used to score each lesion . Before every scoring session, the device was calibrated using the standard ceramic according to the manufacturer's instructions. The teeth were rinsed and air dried before registration and a type B probe tip was positioned on the buccal surface of the tooth and rotated around its vertical axis until the peak reading was displayed on the panel. All measurements were taken 3 times and the average fluorescence value was recorded. Higher DIAGNOdent Pen values indicate deeper caries and the difference between the values obtained at different time intervals and the initial value indicates the amount of change in the loss of fluorescence of the lesions

CONTACTS AND LOCATIONS:
Locations (1):
- Emel Karaman, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richter AE, Arruda AO, Peters MC, Sohn W. Incidence of caries lesions among patients treated with comprehensive orthodontics. Am J Orthod Dentofacial Orthop. 2011 May;139(5):657-64. doi: 10.1016/j.ajodo.2009.06.037. PMID 21536209
- [Background] Tufekci E, Dixon JS, Gunsolley JC, Lindauer SJ. Prevalence of white spot lesions during orthodontic treatment with fixed appliances. Angle Orthod. 2011 Mar;81(2):206-10. doi: 10.2319/051710-262.1. PMID 21208070
- [Background] Ogaard B. Prevalence of white spot lesions in 19-year-olds: a study on untreated and orthodontically treated persons 5 years after treatment. Am J Orthod Dentofacial Orthop. 1989 Nov;96(5):423-7. doi: 10.1016/0889-5406(89)90327-2. PMID 2816842
- [Background] Bergstrand F, Twetman S. A review on prevention and treatment of post-orthodontic white spot lesions - evidence-based methods and emerging technologies. Open Dent J. 2011;5:158-62. doi: 10.2174/1874210601105010158. Epub 2011 Sep 16. PMID 21966335
- [Background] Dogra S, Goyal V, Gupta A, Joshi S, Kataria V, Saini J, Nagpal M, Narula P. Spectrophotometric Evaluation of Color Change in Tooth Enamel Defects Using Resin Infiltrate: An In Vivo Study. Int J Clin Pediatr Dent. 2020 Mar-Apr;13(2):150-154. doi: 10.5005/jp-journals-10005-1727. PMID 32742092
- [Background] Faghihian R, Shirani M, Tarrahi MJ, Zakizade M. Efficacy of the Resin Infiltration Technique in Preventing Initial Caries Progression: A Systematic Review and Meta-Analysis. Pediatr Dent. 2019 Mar 15;41(2):88-94. PMID 30992105
- [Background] Neuhaus KW, Graf M, Lussi A, Katsaros C. Late infiltration of post-orthodontic white spot lesions. J Orofac Orthop. 2010 Nov;71(6):442-7. doi: 10.1007/s00056-010-1038-0. Epub 2010 Nov 17. English, German. PMID 21082307
- [Background] Patcas R, Zinelis S, Eliades G, Eliades T. Surface and interfacial analysis of sandblasted and acid-etched enamel for bonding orthodontic adhesives. Am J Orthod Dentofacial Orthop. 2015 Apr;147(4 Suppl):S64-75. doi: 10.1016/j.ajodo.2015.01.014. PMID 25836346
- [Background] Youssef A, Farid M, Zayed M, Lynch E, Alam MK, Kielbassa AM. Improving oral health: a short-term split-mouth randomized clinical trial revealing the superiority of resin infiltration over remineralization of white spot lesions. Quintessence Int. 2020;51(9):696-709. doi: 10.3290/j.qi.a45104. PMID 32901234